CLINICAL TRIAL: NCT07188129
Title: Assessing Compatibility of the ZywieAI Algorithm to Analyze ECG Data Collected From the Zywiez3 Sensor and Adhesive Over a 24-hour Period
Brief Title: Evaluation of a Test Algorithm for Use to Analyze ECG Data Collected From a Test Device of a 24-hour Simulated Use Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zywie, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2410003-150
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Tachycardia; Bradycardia; PVC - Premature Ventricular Contraction; Premature Atrial Contraction
Keywords: ECG Evaluation Algorithm; Simulated ECG Use
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia; Bradycardia; Ventricular Premature Complexes; Atrial Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Evaluation of 24-hour ECG Data from Test Device by a Test Analysis Algorithm (Other): ECG data will be collected from subjects with previously diagnosed heart arrhythmias by a test algorithm. ECG data collected using a Test Device with non-traditional lead placement worn for a 24-hour period. The Test Algorithm analysis will be compared to assessments of the ECG data by 2 cardiologists with a 3rd cardiologist employed when there is no agreement by the 2 cardiologists.
  Interventions: Device: Test Algorithm and Test Device

INTERVENTIONS:
Device: Test Algorithm and Test Device — Test Algorithm analysis of 24-hour ECG Data collected with a Test Device

SUMMARY:
The purpose of this study is to demonstrate that the ZywieAI analysis algorithm can be used to analyze ECG data collected from ZywieZ3 devices with non-traditional lead placement over a 24-hour simulated use period by human subjects.

DETAILED DESCRIPTION:
At least 150 subjects will participate in this study over a 24-hour test period. The subjects must have been diagnosed with a known condition such as Atrial Fibrillation (AF), Tachycardia, Bradycardia, Premature Ventricular Contractions (PVC/VEB), and/or Premature Atrial Contractions (PAC), etc.

A Testing Facility analyst will conduct an initial visual evaluation of the level of skin adhesion for the Test Device. The Testing Facility analyst will apply the Test device adhesive on the subject and initiate ECG data collection. Subjects will observe a 5-minute stabilization period to ensure the device is connected appropriately and has a stable input signal. Subjects will be allowed to leave the Testing Facility for the next 24 hours. During this period, subjects will follow the instructions for use provided by the Sponsor and engage in normal routine activities. After the 24-hour recording, subjects will return to the Testing Facility, and an analyst will then remove the Test Device.

Two cardiologists will review the collected ECG data from the 24-hour wear time to identify episodes of arrhythmia. A third cardiologist will be used to review the ECG data collected if the first two do not agree with their assessment. The Sponsor will download the ECG data for the Test Device from a cloud-based data repository to complete the data analysis according to the Sponsor's statistical analysis plan. The cardiologist's assessment will be compared with the analysis by the ZywieAI algorithm. A summary of the ECG statistical analysis comparing the agreement of the cardiologists will be included as an appendix to the final report for the study.

ELIGIBILITY:
Inclusion Criteria:

* Of the 150 subjects who complete the study, at least 60 (i.e., ≥ 40%) subjects must be male, and at least 60 (i.e., ≥ 40%) subjects must be female.
* Subjects must be more than 18 years of age.
* Subjects' body mass index (BMI) will be calculated based on their weight and height at the time of consent. BMI will be calculated using the CDC's online Adult BMI Calculator (https://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/english_bmi_calculator/bmi_calculator.html). This calculator will also automatically categorize the calculated BMI as underweight to healthy (< 18.5 to 24.9), overweight (25.0 to 29.9), or obese (≥ 30.0). Of the 150 subjects who complete the study, no more than 70 subjects can be from a given BMI category.
* Subjects must be able to read, write, and understand English.
* Subjects must be in good general health (i.e., no current or recent severe illness).
* Subjects must have a known condition of Atrial Fibrillation (AF), Tachycardia, Bradycardia, Premature Ventricular Contractions (PVC/VEB), and/or Premature Atrial Contractions (PAC) diagnosed by a medical professional.
* Subjects with body hair on their upper-left chest must be willing to have the body hair clipped by a Testing Facility analyst before applying the Test Device.
* Subjects must be willing to have their upper-left chest cleaned with 70% isopropanol preparation pads before applying the Test Device.

Exclusion Criteria:

* Subjects cannot be currently participating in another clinical study.
* Subjects cannot have active skin rashes, dermatoses, or breaks in the skin on the upper left chest region.
* Subjects cannot have undergone any surgeries during the last 3 months involving incisions along their upper-left chest.
* Subjects cannot have any tattoos on their upper-left chest.
* Subjects cannot have currently active inflammatory skin conditions (e.g., atopic dermatitis/eczema, contact dermatitis, or psoriasis) anywhere on the body within 2 days of the start of the test period and during the 24-hour test period.
* Subjects cannot have a medical diagnosis of an organ transplant, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an immunocompromised condition such as AIDS (or HIV positive), lupus, medicated fibromyalgia, ulcerative colitis, Crohn's disease, moderate to severe asthma (requiring daily use of medication), or medicated multiple sclerosis.
* Subjects cannot have a pacemaker.
* Subjects cannot have any type of port, shunt, or Peripherally Inserted Central Catheter (PICC).
* Subjects cannot receive any vaccinations within 7 days of the start of the test period and while participating in the 24-hour test period.
* Subjects cannot have known allergies or sensitivities to latex (natural rubber), adhesives, inks, sunscreens, deodorants, laundry detergents, cleansers, soaps, lotions, to topical application of fragrances (e.g., perfumes or colognes), acrylic, hydrogel, isopropyl alcohol, C11-12 isoparaffin, isopropyl palmitate, isopropyl myristate, or isopropyl stearate.
* Subjects cannot be pregnant, plan to become pregnant, or cause a partner to become pregnant during the study.
* Subjects cannot be nursing a child during the 24-hour test period.
* Subjects cannot have any medical condition or use any medications that, in the opinion of the Principal Investigator or Consulting Physicians, should preclude participation or might impact data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Demonstration that the ZywieAI analysis algorithm can be used to analyze ECG data collected from ZywieZ3 devices with non-traditional lead placement over a 24-hour simulated use period by human subjects | 24 Hours after Application of Test Device
  Two cardiologists will review the collected ECG data from the 24-hour wear time to identify episodes of arrhythmia. A third cardiologist will be used to review the ECG data collected if the first two do not agree with their assessment. The Sponsor will download the ECG data for the Test Device from a cloud-based data repository to complete the data analysis by ZywieAI algorithm identifying cardiac anomalies. The cardiologist's assessment will be compared with the analysis by the ZywieAI.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Beausoleil, B.S., Principal Investigator — Bioscience of Bozeman LLC
Locations (1):
- Bioscience of Bozeman, LLC, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans for publishing the data from this trial.